CLINICAL TRIAL: NCT01736709
Title: A Single-centered, Open-labeled, Phase 4 Study of 2012-2013 Trivalent Seasonal Influenza Vaccine
Brief Title: The Immunogenicity and Safety of 2012-2013 Trivalent Seasonal Influenza Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO-INF-4012
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2012-11

CONDITIONS: Influenza
Keywords: 2012-2013 trivalent seasonal influenza vaccine; immunogenicity,; safety
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- trivalent seasonal influenza vaccine (Experimental): 2012-2013 trivalent seasonal influenza vaccine in 60 infants with two-dose regimen, 21 days interval trivalent seasonal influenza vaccine in 60 adults and 60 old people with single-dose regimen
  Interventions: Biological: 2012-2013 trivalent seasonal influenza vaccine

INTERVENTIONS:
Biological: 2012-2013 trivalent seasonal influenza vaccine — trivalent seasonal influenza vaccine with 0.25 ml ⁄ vial, for infants trivalent seasonal influenza vaccine with 0.5 ml ⁄ vial, for adults and old people

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of 2012-2013 trivalent seasonal influenza vaccine in 60 healthy infants aged 6-35 months old, 60 healthy adults aged 18-60 years old, and 60 healthy older people aged > 60 years.

ELIGIBILITY:
For adults and old people:

Inclusion Criteria:

* Healthy adults aged 18-60 years old, and healthy old people aged >60 years
* Be able to show legal identity card for the sake of recruitment Without vaccination history of seasonal split influenza vaccine in the recent 3 years
* Not participate in any other clinical trials during the study
* Not receive any immunosuppressive agents during and one month prior to the study
* Be able to understand and sign the informed consent.

Exclusion Criteria:

* Woman： Who breast-feeding or planning to become pregnant during the study
* Any history of allergic reactions; was allergic to any component of the vaccine, such as eggs or ovalbumin
* Any history of severe adverse reactions to vaccines, such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Acute episode of chronic diseases or conditions, including chronic hepatitis, hypertension, diabetes mellitus and cardiovascular diseases
* Guillain-Barre Syndrome
* Women subjects with positive urinary pregnancy test
* Any history of immunosuppressive medications or cytotoxic medications or inhaled corticosteroids within the past six months (with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis)
* Axillary temperature >37.0 centigrade at the time of dosing
* Psychiatric condition that precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder requiring therapy that has not been well controlled on medication for the past two years; disorder requiring lithium; or suicidal ideation occurring within five years prior to enrollment
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent.

For infants:

Inclusion Criteria:

* Healthy male or female aged between 6 and 35 months
* Full-term birth, birth weight 2,500 grams or more
* provided birth certification or vaccination card Parent(s) or legal guardian(s) are able to understand and sign the informed consent

Exclusion Criteria:

* Administration of 2012-2013 seasonal vaccine
* Subject that has a medical history of any of the following: allergic history, or allergic to any ingredient of vaccine, such as egg, egg protein, etc
* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Symptoms of acute infection within a week
* Autoimmune disease or immunodeficiency
* Congenital malformation, developmental disorders or serious chronic diseases (such as Down's syndrome, diabetes, sickle cell anemia or neurological disorders)
* Asthma that is unstable or required emergent care, hospitalization or intubation during the past two years or that required the use of oral or intravenous corticosteroids
* Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with Intramuscular injections or blood draws
* History or family history of convulsions, epilepsy, brain disease and psychiatric
* Asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen
* Guillain-Barre Syndrome
* History of any blood products within 3 months
* Administration of any other investigational research agents within 30 days
* Administration of any live attenuated vaccine within 30 days
* Administration of subunit or inactivated vaccines within 14 days
* Be receiving anti-Tuberculosis prophylaxis or therapy currently
* Axillary temperature > 37.0 centigrade at the time of dosing
* Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer's ability to give informed consent

Ages: 6 Months to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-11; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Hemagglutination inhibition (HI) antibody titer of 2012-2013 trivalent seasonal influenza vaccine | 21 days after vaccination
  to evaluate the immunogenicity of the vaccine in adults and old people.

SECONDARY OUTCOMES:
Frequency of systemic and local adverse reactions after vaccination | 0-21 days after vaccination
  to evaluate the safety of the vaccine in healthy infants, adults, and old people

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Shen Guo, BS, Principal Investigator — Henan Center for Diseases Control and Prevention
Locations (1):
- Henan Center for Diseases Control and Prevention, Zhengzhou, Henan, China